CLINICAL TRIAL: NCT05524623
Title: Comparative Effect of Percutaneous Microelectrolysis With or Without Current Emission in the Treatment of Cervical Pain in Myofascial Trigger Points of the Trapezius
Brief Title: Comparative Effect of MEP With or Without Current Emission in the Treatment of Cervical Pain in MTrPs of the Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, Arguello Retamar Verónica Inés, Principal Investigator (Bachelor of Kinesiology and Physiotherapy), Universidad Nacional de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3926
Record Dates: First submitted 2022-08-13; First posted 2022-09-01 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Neck Pain, Posterior; Myofascial Pain Syndromes
Keywords: neck; pain; muscles; needles; Electrolysis; electrotherapy
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes; Pain

STUDY DESIGN:
Intervention Model Description: percutaneous microelectrolysis with or without current emission in the treatment of cervical pain in myofascial trigger points of the trapezius. Both will take place over 3 weeks, with one session per week. The evaluation is carried out through the visual analogue scale (VAS), measurement of force with a dynamometer and mobility with a goniometer. The score will be recorded on a validated neck pain questionnaire (NPQ).
Who Masked: Participant
Masking Description: Both groups do not know if the treatment has emission or not while the sessions are carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without current emission in the treatment (Sham Comparator): percutaneous microelectrolysis without current emission in the treatment of cervical pain in myofascial trigger points of the trapezius. Both will take place over 3 weeks, with one session per week.
  Interventions: Other: percutaneous microelectrolysis in myofascial trigger points of the trapezius
- wit current emission in the treatment (Active Comparator): percutaneous microelectrolysis with current emission in the treatment of cervical pain in myofascial trigger points of the trapezius. oth will take place over 3 weeks, with one session per week.
  Interventions: Other: percutaneous microelectrolysis in myofascial trigger points of the trapezius

INTERVENTIONS:
Other: percutaneous microelectrolysis in myofascial trigger points of the trapezius — percutaneous microelectrolysis with or without current emission in the treatment of cervical pain in myofascial trigger points of the trapezius
  Other Names: MEP (percutaneous microelectrolysis); Trigger Points

SUMMARY:
Myofascial pain syndrome (MPS) is initial to other pathologies such as neck pain or tension headaches; the symptoms that are located on the area of myofascial trigger points (MTrPs) of specific references in different muscles. MTrPs are palpable, tense bands found in stiff muscle that cause pain and swelling. They affect the disruptive soft tissues, resulting in deterioration of the muscle and fascia; effects that can be transferred further, through the myofascial chain to distant tissues, inducing the referred pain that is the main feature of MPS. MTrPs are treated with stretching, massage, analgesics, acupuncture, dry needling, electrical stimulation, and ultrasound. Percutaneous microelectrolysis (MEP®) is a new technique that uses galvanic current of low intensity and high density. Based on the previous reviews, the investigators consider that the use of MEP in individuals who have MTrPs in the trapezius is more effective than acupuncture treatment. Objectives: To assess the effect of MEP as a technique for treating pain in MTrPs of the trapezius muscle compared to without current emission, analyzing function, pain and strength in MTrPs before and after both treatments.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is initial to other pathologies such as neck pain or tension headaches; the symptoms that are located on the area of myofascial trigger points (MTrPs) of specific references in different muscles. MTrPs are palpable, tense bands found in stiff muscle that cause pain and swelling. They affect the disruptive soft tissues, resulting in deterioration of the muscle and fascia; effects that can be transferred further, through the myofascial chain to distant tissues, inducing the referred pain that is the main feature of MPS. MTrPs are treated with stretching, massage, analgesics, acupuncture, dry needling, electrical stimulation, and ultrasound. Percutaneous microelectrolysis (MEP®) is a new technique that uses galvanic current of low intensity and high density. Based on the previous reviews, the investigators consider that the use of MEP in individuals who have MTrPs in the trapezius is more effective than acupuncture treatment. Objectives: To assess the effect of MEP as a technique for treating pain in MTrPs of the trapezius muscle compared to without current emission, analyzing function, pain and strength in MTrPs before and after both treatments.

Materials and methods: Randomized controlled clinical research. The study population consists of patients of both sexes between 20 and 60 years of age, with medical referral for neck pain who do not currently receive physiotherapeutic treatment, pain of at least 1 month of evolution, presenting on both sides of the trapezius MTrPs muscle and having signed the informed consent. They will be randomly distributed into: group treated with acupuncture (control) and group treated with MEP. Both will take place over 3 weeks, with one session per week. The evaluation is carried out through the visual analogue scale (VAS), measurement of force with a dynamometer and mobility with a goniometer. The score will be recorded on a validated neck pain questionnaire (NPQ). The Chi-Square test (test) will be implemented for the analysis of categorical data and the "t" test for paired data for quantitative data, based on a significance level of p˂0.05 in all cases.

ELIGIBILITY:
Inclusion Criteria:

* with medical referral for pain of at least 1 month of evolution
* presenting on both sides of the trapezius MTrPs muscle

Exclusion Criteria:

* neck pain who do currently receive physiotherapeutic treatment of at least 1 month of evolution

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Northwick Park Neck Pain Questionnaire | will take place over 3 weeks, with one session per week.
  The validated and adapted Northwick Park Neck Pain Questionnaire (NPQ) relates to activities of daily living. The outcome measure is in Points per NPQ protocol. The questionnaire will be completed prior to treatment. Nominal variables were described by of proportions with a confidence interval of 95%; Chi-Square test (Pearson's test), based on a significance level of p˂0.05 in all cases.
Mobility with a goniometer | will take place over 3 weeks, with one session per week.
  The range of joint mobility of flexion, extension, inclination and rotation movements will be measured with a goniometer. The outcome measure is in degrees, before and after treatment. Evaluating the comparative effect of percutaneous microelectrolysis with or without current emission in the treatment of cervical pain in trapezius myofascial trigger points.
Objective pain measurement with a dynamometer | will take place over 3 weeks, with one session per week.
  It is the objective measurement of pain, through the measurement of results in the Newton (N) unit to perform force measurements and objectively evaluate the pain threshold at strategic points of the trapezius muscle, using the DINATOR® portable dynamometer. It will be measured with the dynamometer before and after treatment with or without current. Evaluated comparative effect of percutaneous microelectrolysis with or without current emission in the treatment of cervical pain in myofascial trigger points of the trapezius.
visual analogue scale | will take place over 3 weeks, with one session per week.
  The evaluation is carried out through the visual analogue scale (VAS) with the outcome measure from 0 to 10 (10 the worst pain experienced and 0 no pain); change from pain level to baseline pain level before and after treatment. The Chi-Square test (Pearson's test) will be implemented for the analysis of categorical data and the "t" test for paired data for quantitative data, based on a significance level of p˂0.05 in all cases. Evaluated comparative effect of percutaneous microelectrolysis with or without current emission in the treatment of cervical pain in myofascial trigger points of the trapezius.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Campana, Dr, Study Director — Universidad Nacional de Córdoba
Locations (1):
- Centro de Investigación, Extensión y Capacitación de la Escuela de Kinesiología y Fisioterapia, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Margalef R, Bosque M, Monclus P, Flores P, Minaya-Munoz F, Valera-Garrido F, Santafe MM. Percutaneous Application of Galvanic Current in Rodents Reverses Signs of Myofascial Trigger Points. Evid Based Complement Alternat Med. 2020 May 28;2020:4173218. doi: 10.1155/2020/4173218. eCollection 2020. PMID 32565858
- See also: Percutaneous Application of Galvanic Current in Rodents Reverses Signs of Myofascial Trigger Points — https://pubmed.ncbi.nlm.nih.gov/32565858/

DOCUMENTS (1):
  • Informed Consent Form (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT05524623/ICF_000.pdf